CLINICAL TRIAL: NCT03077373
Title: The Efficacy of a Computerized Brief Intervention Targeting Physical Activity, Sedentary Behavior, and Smoking Cessation on the Reduction of Systolic Blood Pressure in Individuals Aged 40 to 65 Years
Brief Title: Efficacy of a Brief Intervention on Reduction of Systolic Blood Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: BB005/17
Record Dates: First submitted 2017-03-07; First posted 2017-03-10 (Actual); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Blood Pressure, High; Cardiovascular Risk Factor
Keywords: systolic blood pressure; physical activity; sedentary time; smoking
MeSH Terms: conditions — Hypertension; Motor Activity; Sedentary Behavior; Smoking

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Counseling letter (intervention group) (Experimental): Intervention group: Individuals in this group complete a tablet PC-supported assessment at baseline and 12-month follow-up, both at the general practice. At months 4 and 7, follow-up data are collected by study team members via phone call. According to the assessments (baseline, month 4, and month 7), participants receive three counseling letters aiming to increase moderate-to-vigorous physical activity and to reduce sedentary time. Additionally, individuals who were daily smokers at baseline, receive three counseling letters aiming to foster the motivation to quit smoking. The first letter is accompanied by a self-help manual covering specific information relevant for the particular stage of motivation to change smoking behavior.
  Interventions: Behavioral: Counseling letter
- No counseling letter (control group) (No Intervention): Control group: Individuals in this group complete a tablet PC-supported assessment at baseline and 12-month follow-up, both in the general practice. At months 4 and 7, follow-up data are collected by study team members via phone call.

INTERVENTIONS:
Behavioral: Counseling letter — The brief counseling letter intervention aiming to reduce physical inactivity, sedentary time in leisure time as well as smoking is based on behavior change theories (Transtheoretical model of health behavior change and Health Action Process Approach).
  The computerized intervention system includes up to six interactions with participants. Recurrent assessments are initiated by the system and provide data for scheduling the proceeding intervention steps and selection of relevant content. Physical activity, sedentary time, smoking, and motivational measures to change or maintain behaviors according to the recommendations will be monitored over time and used to provide feedback in the form of letters.
  Arms: Counseling letter (intervention group)

SUMMARY:
This study examines the efficacy of individualized counseling letters to reduce systolic blood pressure level of ≥ 130 mmHg in individuals aged between 40 and 65 years. The computer-generated counseling letter intervention aimed to increase moderate-to-vigorous physical activity, to reduce sedentary time, and to achieve smoking abstinence.

DETAILED DESCRIPTION:
This study examines the efficacy of individualized counseling letters to reduce systolic blood pressure level of ≥ 130 mmHg in individuals aged between 40 and 65 years. The computer-generated counseling letter intervention aimed to increase moderate-to-vigorous physical activity, to reduce sedentary time, and to achieve smoking abstinence. Participants are recruited by nurses in routine care of primary medical practices.

Informed consent consists of: (i) participation in standardized measurement of blood pressure as well as waist and hip circumference at baseline and 12-month follow up, (ii) completion of standardized questionnaires at 4 time points (baseline, 4-month, 7-month, and 12-month follow-up). Participation in accelerometry was defined as an option. Individuals who agree to wear the accelerometer do this for 10 days at baseline and 12-month follow-up, each.

After baseline assessment, individuals are randomly allocated to a control and to an intervention group (ratio 1:1).

Intervention: The computerized intervention system includes three interactions with participants aiming to increase moderate-to-vigorous physical activity and to reduce sedentary time. For individuals who were daily smokers at baseline, the computerized intervention system includes three more interactions with participants aiming to foster the motivation to quit smoking. Recurrent assessments are initiated by the system and provide data for scheduling the proceeding intervention steps and selection of relevant content. Physical activity, sedentary time, smoking, and motivational measures to change or maintain behaviors according to the recommendations will be monitored over time and used to provide feedback in the form of letters.

Intervention group: Individuals in this group complete a tablet PC-supported assessment at baseline and 12-month follow-up, both at the general practice. At months 4 and 7, follow-up data are collected by study team members via phone call. According to the assessments (baseline, month 4, and month 7), participants receive three counseling letters aiming to increase moderate-to-vigorous physical activity and to reduce sedentary time. Additionally, individuals who were daily smokers at baseline, receive three counseling letters aiming to foster the motivation to quit smoking. The first letter is accompanied by a self-help manual covering specific information relevant for the particular stage of motivation to change smoking behavior according to the principles of the Transtheoretical Model of behavior change.

Control group: Individuals in this group complete a tablet PC-supported assessment at baseline and 12-month follow-up, both in the general practice. At months 4 and 7, follow-up data are collected by study team members via phone call.

ELIGIBILITY:
Inclusion Criteria:

* men and women aged between 40 and 65 years
* mean systolic blood pressure ≥ 130 mmHg at baseline

Exclusion Criteria:

* cardiovascular event (myocardial infarction, stroke)
* vascular intervention
* cognitive impairment
* inadequate language skills
* severe disease with reduced life expectancy (< 2 years)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure | Change from baseline mean systolic blood pressure at 12 months
  Reduction of 4 mmHg mean systolic blood pressure in intervention group; Measures: standardized measurements of mean systolic blood pressure (in mmHg)

SECONDARY OUTCOMES:
Waist and hip circumference | Change from baseline waist and hip circumference at 12 months
  Reduction of waist and hip circumference in intervention group; Measures: standardized measurements of waist and hip circumference (in cm)
Physical activity by self-report | Change from baseline physical activity at 12 months
  Measures: assessement via tablet PC or phone calls (International Physical Activity Questionnaire, IPAQ)
Physical activity by accelerometry (if data are available) | Change from baseline physical activity at 12 months
  Measures: objective measurement of physical activity by accelerometry
Sedentary time by self-report | Change from baseline sedentary time at 12 months
  Measures: assessement via tablet PC or phone calls (last 7-d sedentary behavior questionnaire, SIT-Q-7d)
Sedentary behavior by accelerometry (if data are available) | Change from baseline physical inactivity at 12 months
  Measures: objective measurement of sedentary behavior by accelerometry
Smoking by self-report | Change from baseline smoking at 12 months
  Measures: questions regarding smoking (assessment via tablet PC or phone calls)

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Ulbricht, Dr., Study Chair — Institute of Social Medicine and Prevention, University Medicine Greifswald, Greifswald, Germany
Locations (1):
- Institute of Social Medicine and Prevention, University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: Undecided